CLINICAL TRIAL: NCT05979961
Title: Concurrent Chemoradiotherapy Alone Versus Induction Chemotherapy Plus Concurrent Chemoradiotherapy in Low-risk Locoregionally Advanced Nasopharyngeal Carcinoma: a Phase 3, Multicentre, Randomised Controlled Trial
Brief Title: Phase III Trial of Concurrent Chemotherapy Alone in Patients With Low-risk Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Tongji Hospital (Other); Guangzhou Panyu Central Hospital (Other); Hunan Cancer Hospital (Other); Cancer Hospital of Guizhou Province (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-FXY-298
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Induction Chemotherapy; Concurrent Chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Gemcitabine; Cisplatin; Induction Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMRT and concurrent cisplatin (Experimental): Patients receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin 100 mg/m² every 3 weeks for 3 cycles.
  Interventions: Radiation: IMRT and concurrent cisplatin
- Induction chemotherapy+IMRT and concurrent cisplatin (Active Comparator): Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 3 cycles before radiotherapy, and then receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin 100 mg/m² every 3 weeks for 3 cycles.
  Interventions: Radiation: IMRT and concurrent cisplatin; Drug: gemcitabine and cisplatin (Induction chemotherapy)

INTERVENTIONS:
Radiation: IMRT and concurrent cisplatin — Patients receive concurrent cisplatin 100mg/m2 every 21days for three cycles during Intensity modulated radiotherapy (IMRT)
Drug: gemcitabine and cisplatin (Induction chemotherapy) — Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for 3 cycles before radiotherapy
  Arms: Induction chemotherapy+IMRT and concurrent cisplatin

SUMMARY:
The purpose of this study is to compare concurrent chemoradiotherapy (CCRT) alone with induction chemotherapy (gemcitabine+cisplatin) plus CCRT in patients with low-risk locoregionally advanced nasopharyngeal carcinoma(NPC).

DETAILED DESCRIPTION:
Patients with low risk NPC( Stage III-IVa, except T4N2/AnyTN3, AJCC 8th and EBV DNA <4000 copies/ml) are randomly assigned to receive CCRT alone or induction chemotherapy plus CCRT. Patients in both groups receive cisplatin 100 mg/m² every 3 weeks for 3 cycles, concurrently with intensity-modulated radiotherapy (IMRT). IMRT is given as 2.12 Gy per fraction with five daily fractions per week to a total dose of 70 Gy. The induction chemotherapy plus CCRT group receive gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for three cycles before CCRT. Our primary endpoint is progress-free survival. Secondary end points include overall survival (OS), Locoregional progression, Distant progression and toxic effects. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old.
2. Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type).
3. Tumor staged as III-IVa except T4N2/AnyTN3 (according to the 8th AJCC edition) and pretreatment plasm EB Virus DNA<4000copies/ml.
4. ECOG Performance status less or equal to 1.
5. Male and no pregnant female.
6. Adequate marrow: leucocyte count ≥ 4000/μL, hemoglobin ≥ 90g/L and platelet count ≥ 100000/μL.
7. Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) < 2.5×ULN, and bilirubin < ULN.
8. Adequate renal function: creatinine clearance ≥ 60 ml/min.
9. Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

1. Patients have evidence of relapse or distant metastasis.
2. WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
3. Treatment with palliative intent.
4. History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume).
5. Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
6. Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
7. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
8. Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival(PFS) | 3 years
  defined as the time from random assignment to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  defined as the time from random assignment to death from any cause.
Locoregional progression | 3 years
  defined as the time from random assignment to the occurrence of a locoregional progression. Cumulative incidence of locoregional progression will be calculated within a competing risk framework (Fine and Gray 1999).
Distant progression | 3 years
  defined as the time from random assignment to the occurrence of a distant progression. Cumulative incidence of distant progression will be calculated within a competing risk framework (Fine and Gray 1999).
Overall response rate | 16 weeks after completion of concurrent chemoradiotherapy
  Tumour response was classified according to RECIST, version 1.1
Incidence of acute and late toxicity | 3 years
  Incidence of acute toxicity is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Cancer Hospital of Guizhou Province, Guiyang, Guizhou
  - Tongji Hospital,Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College,Huazhong University of Science and Technology;, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan